CLINICAL TRIAL: NCT04971538
Title: Cluster Randomized Controlled Study of Home-based Hepatitis C Self-testing in Karachi, Pakistan
Brief Title: HCV Self-testing in Pakistan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HC023
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Hepatitis C; Diagnostic Self Evaluation
Keywords: self-test; micro-elimination; house to house screening
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: This study is a matched cluster randomized controlled study, the households in the intervention clusters will be left information on the importance of testing, an HCV self-test and instructions for use while the households in the control clusters will be left information on the importance of testing for HCV and information on how to get tested at the nearest facility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCV self-testing (Experimental): the study staff will leave an HCV ST and instructions for use (IFU) with the household. The study team will also explain the HCVST process to the most senior member of the household, as well as leave a mobile number for the participant to contact for help conducting the test. The study team will follow up with the participant to inquire about if testing was completed, collect any testing results, and conduct a brief survey.
  Interventions: Diagnostic Test: OraQuick® HCV Self-Test
- Referral to clinic for HCV RDT (No Intervention): the study staff will leave information on HCV testing and direct them to the nearest clinic with screening services, the participant will not be left a HCVST. Study staff will also leave a mobile number for the participant to contact for further information on HCV testing. The study team will follow up with the participant to inquire about if testing was completed, collect any testing results, and conduct a brief survey

INTERVENTIONS:
Diagnostic Test: OraQuick® HCV Self-Test — The OraQuick® HCV Self-Test is a lateral flow rapid diagnostic that can detect anti-HCV antibodies in oral fluid. Instructions for Use (IFU) for OraQuick® HCV Rapid Antibody Self-Test have been developed in Georgian for the previous 2 studies conducted in Georgia using the OraQuick® HCV Rapid Antibody Self-Test. The IFU has been optimized taking in the feedback on the IFU resulting from the aforementioned studies. As this HCV test is not approved for self-test use in Georgia, all tests will be labelled as Research Use Only (RUO) and test results will not be used for patient management.
  Arms: HCV self-testing

SUMMARY:
To achieve the goal of elimination of hepatitis C infection in Pakistan, the strategy of elimination needs to be increasingly directed towards case finding through mass screening in rural or peri-urban communities to identify and treat those not yet aware of their infection.

Self-testing (ST) with easy-to-use rapid diagnostic tests has been successfully used for diseases such as HIV. The availability of self-testing has been shown to increase testing rates and testing acceptability in diverse populations around the world, in large part due to its convenience and privacy advantages. In the present study we aim to evaluate the acceptability and impact of a program enabling home delivery of hepatitis C virus (HCV) self-testing in the Malir district, Karachi division, Pakistan.

DETAILED DESCRIPTION:
This study is a cluster randomized controlled study that will be nested within a larger micro-elimination study run by Aga Khan University (AKU). This larger study has already completed house-to-house screening of Union Council (UC) 9 and 10 in the Malir district of Karachi, with a number of households still in need of follow-up, these households contained members who were not present during the house-to-house screening and were not able to be offered the HCV rapid diagnostic test (RDT). In this study AKU study staff will return to the households that had persons missed by the first round of house-to-house screening done during the CHIME study.

For randomization purposes, the neighborhoods in UC 9 and 10 will be grouped into clusters. The clusters will be matched in pairs based on similarity of geography (peri-urban or rural), population size, and age demographics. Each cluster within a matched pair will then be randomized to the intervention or control group.

In the intervention group, if the participant is not home the study staff will leave an HCV self test (HCV ST), instructions for use ( IFU), and supporting materials with the household. The study team will also explain the HCVST process to the most senior member of the household, as well as leave a mobile number for the participant to contact for help conducting the test. The study team will follow up with the participant to inquire about if testing was completed. If the HCV ST is reactive, study staff, over the phone, will also make an appointment to return to the house for enrolment into the larger AKU micro-elimination study, and after enrolment into the lager AKU micro-elimination study the participant will receive a blood draw for HCV RNA confirmatory testing and APRI staging. If the participant is HCV viraemic they will be provided treatment, delivered to their door by The Liver Foundation.

In the control group, if the participant is not home the study staff will leave both printed and verbal information on HCV testing and direct them to the nearest clinic with screening services. Study staff will also leave a mobile number for the participant to contact for further information on HCV testing. The study team will follow up with the participant to inquire about if testing was completed. If the HCV test is reactive, study staff, over the phone, will also make an appointment to return to the house for enrolment into the larger AKU micro-elimination study, and after enrolment into the lager AKU micro-elimination study the participant will receive a blood draw for HCV RNA confirmatory testing and Aspartate aminotransferase to Platelet Ratio Index (APRI) staging. If the participant is HCV viraemic they will be provided treatment, delivered to their door by The Liver Foundation.

In both groups result reporting of did the test and it was positive, did the test and it was negative and did the test and it was indeterminate/I don't know the result, and did not do the test will be incentivized with a 500-rupee phone credit voucher, for those participants who phone AKU and inform them of the results within one month of enrolment. The study team will follow up with a subsection of participants, n=60 in the intervention and n=60 in the control, conduct a brief survey on their perceptions of the testing process

In both groups, if the previously missed person is home when the study staff visits, that person will be enrolled in the larger micro-elimination study and not this study, no self-testing will be done. Study staff will conduct onsite RDT testing and reflex blood draw for confirmatory HCV RNA testing and APRI staging if the RDT is reactive as per the larger study protocol. If the person has HCV viremia, they will be provided HCV tx delivered to their door by The Liver Foundation.

An operational analysis and a costing analysis will also be done evaluating the costs associated with self-testing home delivery with regards to cost per test completed and cost per person diagnosed with HCV.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Residing in UC 9 or 10
* Eligible for inclusion in the larger AKU micro-elimination study

Exclusion Criteria:

* Known to be HCV antibody positive
* Tested for HCV within the last 6 months
* At home during the visit by AKU staff for this study and available to be tested by study staff with an onsite RDT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of HCV self-testing home delivery on HCV antibody testing rates | 2 weeks to 2 months after enrollment
  The number of participants who report completing the HCV antibody testing in the intervention group.
To assess the impact of HCV self-testing home delivery on HCV antibody testing rates | 2 weeks to 2 months after enrollment
  To assess that the proportion of participants who report completing the HCV antibody testing in the intervention group is superior to that of the participants in the control group by a margin of 20%.

SECONDARY OUTCOMES:
To assess the impact of HCV self-testing on the number of HCV antibody positive individuals who are aware of their status | 2 weeks to 2 months after enrollment
  Number of HCV antibody positive participants made aware of their status in the intervention vs control group
To assess the cost of HCV self-testing | entire duration of study, estimated 6 months
  Cost per test completed, cost per person diagnosed (serology, RNA) in the intervention vs control groups. The costs of each step on the testing pathway will be combined to determine the overall cost per person diagnosed with HCV viremia

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Hamid, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shilton S, Ali D, Hasnain A, Abid A, Markby J, Jamil MS, Luhmann N, Nabeta P, Ongarello S, Reipold EI, Hamid S. Protocol for a cluster randomised controlled trial of secondary distribution of hepatitis C self-testing within the context of a house-to-house hepatitis C micro-elimination programme in Karachi, Pakistan. BMC Public Health. 2022 Apr 9;22(1):696. doi: 10.1186/s12889-022-13125-9. PMID 35397544